CLINICAL TRIAL: NCT02620059
Title: Development and Evaluation of a Lifestyle Intervention Program for Women' Weight Reduction After Childbirth
Brief Title: A Lifestyle Program on Healthy Weight in Postpartum Period
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IR.TUMS.REC.1394.485
Record Dates: First submitted 2015-10-19; First posted 2015-12-02 (Estimated); Last update posted 2018-05-01 (Actual); Status verified 2015-12

CONDITIONS: Weight Reduction
Keywords: Postpartum Period
MeSH Terms: conditions — Weight Loss

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lifestyle Intervention (Experimental): Behavioral: Lifestyle Intervention These women will receive the Healthy Lifestyle Intervention. This intervention will have been delivered during 12 weeks, which will be Distance learning program (multimedia or internet). During the intervention (12 weeks) and follow up period, women will receive not only motivational messages through the Short Message System (SMS) but also a pedometer to record their steps.The intervention will focus on women increasing physical activity (walking) to 10'000 steps per day and receiving healthy eating guidelines.
  This intervention curriculum will cover topics related to healthy eating, physical activity, and stress management during postpartum. General information about postpartum period will also be provided.
  Interventions: Behavioral: Lifestyle Intervention
- Control (No Intervention): These women will receive general information via pamphlet about postpartum period and tips for stress management.

INTERVENTIONS:
Behavioral: Lifestyle Intervention — The investigators will provide information on healthy eating and physical activity. They will give pedometers to the participants to monitor their daily steps in order to increase it till 10000 steps/day.
  Arms: Lifestyle Intervention

SUMMARY:
The aim of this study is to examine the impact of lifestyle intervention on postpartum weight loss. So the investigators will have two groups in this study. In Experimental group women will receive the Healthy Lifestyle Intervention. This intervention will have been delivered during 12 weeks. In Control group women will receive general information via pamphlet about postpartum period and tips for stress management.

DETAILED DESCRIPTION:
This study will be conducted in two phases. In the first phase , the investigators will conduct a cross-sectional study to assess factors related to the healthy lifestyle after childbirth based on the PRECEDE model. Regarding results of the study, the investigators will plan and implement a lifestyle promoting intervention and will evaluate the effect of the intervention on weight reduction among postpartum women.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy
* Lactating
* Non-smoking
* Full-term birth
* Lack of medical problems
* Lack of any pregnancy-related complications (eg, multiple pregnancy, fetal anomalies, fetal or maternal complications in current or previous pregnancy, and hypertension in pregnancy).
* Nonparticipation in other studies which may affect the results.
* 18.5≤ BMI≤29 before pregnancy
* Women who are sedentary according to the International Physical Activity Questionnaire.

Exclusion Criteria:

* Unwilling to continue participation in the study
* Pregnancy during the study
* Suffering physical problems during the study
* Smoking after birth

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2017-02-19 (Actual); Study Completion 2017-10-30 (Actual)

PRIMARY OUTCOMES:
Body weight changes | Changes from baseline at 12 months postpartum
  The investigators will assess body weight changes through BMI (kg/m2)

SECONDARY OUTCOMES:
Dietary intake changes | Changes from baseline at 12 months postpartum
  The investigators will assess dietary intake changes with 24 hours dietary recall.
Physical activity changes | Changes from baseline at 12 months postpartum
  The pedometer will measure the number of steps.

OTHER OUTCOMES:
Postpartum weight retention changes | Changes from baseline at 12 months postpartum
  Postpartum weight retention will be measured by calculating the difference between weight at a certain time in the postpartum period and weight before pregnancy using a weight scale.
Stress management changes | Changes from baseline at 12 months postpartum
  Stress will be assessed by the Health Promoting Lifestyle Profile (Adult Version) Scale.
Cognitive changes based on the selected behavior change model/s | Changes from baseline at 12 months postpartum
  Cognitive changes will be assessed through questionnaire developed based on behavior change model/s.

IPD SHARING:
Plan to Share IPD: Undecided